CLINICAL TRIAL: NCT06124222
Title: Prosthetic Rehabilitation and Its Influence on Masticatory Performance and Quality of Life in Patients Treated for Head and Neck Cancer
Brief Title: Prosthetic Rehabilitation and Its Influence on Masticatory Performance and QoL in Patients Treated for HNC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Carlos Moreno Soriano, MSc, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 17/2021
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Quality of Life; Objective Masticatory Performance; Subjective Masticatory Performance; Oral Health
Keywords: Masticatory Performance; Quality of Life; Head Neck Cancer; Oral Rehabilitation
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: * Group A: patients who have not received radiotherapy (RT) in their oncologic treatment (non-irradiated).
  * Group B: patients who have received radiotherapy (RT) in their oncologic treatment (irradiated).
Who Masked: Participant, Investigator
Masking Description: There will be double-blind blinding, since neither the participant nor the principal investigator will be aware of which group (A/B) each patient belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients who have not received RT in their oncologic treatment (non-irradiated).
  Interventions: Procedure: Prosthetic oral rehabilitation
- Group B (Experimental): Patients who have received RT in their oncologic treatment (irradiated).
  Interventions: Procedure: Prosthetic oral rehabilitation

INTERVENTIONS:
Procedure: Prosthetic oral rehabilitation — Prosthetic rehabilitation with fixed and/or removable prosthesis.

SUMMARY:
The main goal of this clinical trial (pilot study) is to evaluate whether prosthetic rehabilitation modifies objective masticatory performance, subjective masticatory performance, quality of life, salivary flow and pH in patients treated for head and neck cancer before and after the placement of fixed and/or removable prostheses.

Hypothesis Prosthetic rehabilitation with fixed and/or removable prostheses modifies objective masticatory performance, subjective masticatory performance, quality of life, salivary flow and pH in non-irradiated patients treated for head and neck cancer compared to irradiated patients.

Study population The study population will consist of patients treated for head and neck cancer who are candidates for prosthetic rehabilitation. The type of prosthetic treatment recommended will be determined by a dental expert in the treatment of these patients.

Interventions

1. - First session and recruitment:

   * Oral health status.
   * Sialometry and salivary pH.
   * Subjective masticatory performance.
   * Objective masticatory performance.
   * Quality of life.
2. - Prosthodontic treatment.
3. - Second session (after insertion of the prosthesis)

   After an adaptation period of ± 15-30 days from the insertion of the prosthesis, the recordings carried out in the first session will be performed again:
   * Oral health status.
   * Sialometry and salivary pH.
   * Subjective masticatory performance.
   * Objective masticatory performance.
   * Quality of life.
4. - Third session (follow-up 6 months)

After a period of time of 3 months ± 7 days after the second session, the recordings carried out in the first and second sessions will be performed again:

* Oral health status.
* Sialometry and salivary pH.
* Subjective masticatory performance.
* Objective masticatory performance.
* Quality of life.

DETAILED DESCRIPTION:
The adverse effects of oncological treatment can alter both the functional and esthetic capabilities of patients, resulting in a diminished quality of life. Dental rehabilitation with prostheses is used to restore the loss of these parameters. Therefore, it is important to know whether patients treated for head and neck cancer improve their masticatory performance, and therefore their quality of life, when rehabilitated with fixed or removable prostheses.

Masticatory function is altered after oncologic treatment in patients with head and neck cancer, causing a decrease in their quality of life. Therefore, there is a need to know whether patients treated for head and neck cancer improve their masticatory performance and masticatory function, and therefore their quality of life, when rehabilitated with fixed or removable prostheses, as well as to know whether this variation in parameters is maintained over time. In addition, it is important to evaluate other aspects that are also directly related to quality of life and masticatory function, such as oral health, the level of salivary secretion and its pH.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age who accept the conditions of the study.
* Patients diagnosed and treated for head and neck cancer in the stable phase of their oncologic pathology.
* Patients in need of prosthetic rehabilitation treatment and who agree to be treated.

Exclusion Criteria:

* Subjects under 18 years of age and/or who do not accept the conditions of the study.
* Diagnosis of cancer in regions other than those mentioned in the inclusion criteria.
* Present a tumor recurrence at the time of the study, undefined oncologic evolutionary situation or under oncologic treatment.
* Presence of orofacial pain or craniomandibular dysfunction hindering mandibular movement and or participation in the study.
* Present a disability to complete the different records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective Masticatory Performance | 6 months
  The chewing test consists of chewing a latex bag with 2g of silicone during 20 chewing cycles counted by the same subject. It will be repeated 5 times. Until 10 grams of Opto-Zeta silicone have been chewed, the masticatory performance will be calculated by median particle size (MPS).
Quality of life | 6 months
  It will be analyzed on the basis of the adapted OHIP-14Sp (Oral Health Impact Profile) questionnaire, which will be given to the patients and completed by them. It consists of 14 questions, grouped in pairs and distributed in the following seven categories: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap.
Subjective masticatory performance | 6 months
  It will be analyzed on the basis of the adapted QMF (Quality of Masticatory Function) questionnaire, which will be given to the patients and completed by them. It consists of 29 questions related to the frequency and ease of chewing different types of food. The questions are classified into five groups: eating and chewing skills, habits, meats, fruits and vegetables.
Sialometry and salivary pH | 6 months
  ▪ Unstimulated salivary secretion: the patient will be seated with the head forward, facilitating the accumulation of saliva on the floor of the mouth. The saliva will be deposited in short intervals in a glass for 5 minutes. The collected content is then measured in a graduated tube. ▪ Stimulated salivary secretion: in the same position as the previous test, the patient will chew a portion of paraffin wax for 5 minutes. Saliva is collected in the glass at short intervals during the chewing period. Afterwards, the content will be measured in a graduated tube. ▪ pH: in one of the vessels with accumulated saliva from the previous tests, the salivary pH will be measured by means of paper strips, whose color will be compared with a visual scale. The color obtained on the strip will be compared with the color scale, which establishes a color for each pH value (1 to 14).

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Moreno Soriano, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No